# TITLE: Prospective, Single-Blinded, Randomized-Controlled Trial Comparing the Performance Profiles of Two Non-Cross-Linked Porcine Dermal Matrices in Abdominal Wall Reconstruction

Statistical Analysis Document Date: February 18, 2025 NCT # NCT02228889

Principal investigator: Jeffrey E. Janis, MD, FACS (Professor of Plastic Surgery)

# Comparative Outcomes of Strattice vs. XenMatrix in Complex Abdominal Wall Reconstruction, PI: Jeffrey Janis, MD

# Molly A. Olson, MS

Updated: 18 February, 2025

# **Contents**

| Statistical Analysis Plan | |
|---|---|
| Overview | |
| Statistical Analysis | |
| Descriptive Analysis | |
| Primary Outcome Analysis | |
| Statistical and Study Design Considerations | |
| Rationale for Combining RCT and Observational Study Data | |
| Choice of Statistical Methods | |
| Methodology implementation notes | |
| Additional comments | |
| References | |
| Additional Exclusion Criteria | 4 |
| | _ |
| Tables | |
| Baseline Characteristics | |
| Surgical Characteristics | |
| 6-week Outcomes | |
| Results | 1( |
| Executive Summary | |
| J . | |
| Unadjusted Random Effects Meta-Analysis (Simple Logistic Regression): | 11 |
| Adjusted Random Effects Meta-Analysis (Multivariable Logistic Regression): | |
| Random Effects Meta-Analysis: Simple Logistic Regression | |
| Forest Plot: Log Odds Scale | 1 |
| Random Effects Meta-Analysis: Multivariable logistic regression | |
| Log Odds Scale | |
| Odds Scale | 1' |
| FAQ | 14 |
| ~~~% | |

# Statistical Analysis Plan

#### Overview

This study aims to evaluate the effect of using XenMatrix or Strattice mesh on the occurrence of surgical site occurrences (SSO) within six weeks post-surgery. Patient-level data were drawn from two sources:

- A single-site randomized controlled trial (RCT), and
- A single-site observational study.

These datasets were combined using a random-effects meta-analysis to generate an overall estimate of the treatment effect of mesh type on the risk of SSO.

## Statistical Analysis

#### **Descriptive Analysis**

An unadjusted analysis comparing mesh was performed.

- Baseline Characteristics: Descriptive statistics (e.g., means or medians for continuous data, counts and proportions for categorical data) were generated for both the RCT and observational cohorts.
- Group Comparisons:
  - Continuous variables were compared using the Kruskal-Wallis test.
  - Categorical variables were compared using Pearson's Chi-square test.

#### Primary Outcome Analysis

SSO within 6 weeks was analyzed using logistic regression. Separate logistic regression models were fit for the RCT and for the observational cohort, with mesh type (XenMatrix vs. Strattice) as the primary predictor. Simple logistic regression and multivariable logistic regression was used for each study type (RCT and observational). Both models were adjusted by hernia width, CDC wound class, immunosuppression, and recurrent hernia to account for potential confounding in the observational group. Covariates were selected based on evidence in the literature as well as potential imbalance. The final number of covariates was limited to avoid model overfitting.

#### Confounders:

- Hernia width
- Wound class
- Immunosuppression
- Recurrent hernia

After obtaining separate estimates from the RCT and observational cohort, a random-effects meta-analysis was performed to derive a combined estimate. A combined estimate for the log odds ratio was calculated using inverse variance weighting and a restricted maximum likelihood estimator. Between-study heterogeneity was assessed by the  $I^2$  measure.

Forest plots and summary tables for the log odds ratio and odds ratio were generated to summarize results.

# Statistical and Study Design Considerations

### Rationale for Combining RCT and Observational Study Data

- RCT was terminated early for difficulties with enrollment, resulting in very imbalanced group sizes.
- While some guidelines caution against combining observational studies with RCTs in a single meta-analysis due to methodological differences [2], other sources emphasize that in many situations, the benefits of incorporating all available evidence can outweigh the drawbacks, provided proper methods are used [2, 3]
- [3] proves a framework for synthesis of non-randomized and randomized studies.
  - In this study, the observational data come from the same single site as the RCT and are not subject to publication bias.

#### Choice of Statistical Methods

- Frequentist methods were chosen for broader audience familiarity. Although Bayesian multi-level models are an option, they can be sensitive to prior specification, and the intended audience may be less familiar with them.
- There are not enough events to perform analysis for other outcomes.
- Propensity score matching was not used because it can substantially reduce the sample size (i.e., discarding unmatched patients).

- Statistical methods chosen to maximize data (Propensity score matching methods throw away data). Methods were also chosen based on what audiences would be most familiar with (Frequentist approaches). Bayesian multi-level models are also a choice, but audiences are not as familiar with them and they can be sensitive to priors. as well as
- Because the study was stopped due to practice changes, interpreting results from an early stopped trial can be complex due to potential bias.
- The RCT power calculation is not valid when adding observational data to "boost" sample size, because the assumptions behind RCT power calculations (particularly randomization and control over selection) do not apply to non-randomized data.
- Here is an example of a study using the same methods: Varges D, Manthey H, Heinemann U, et alDoxycycline in early CJD: a double-blinded randomised phase II and observational studyJournal of Neurology, Neurosurgery & Psychiatry 2017;88:119-125.

#### Methodology implementation notes

• Six patients were missing hernia size; mesh size was used as a proxy in those cases. While not ideal, this approach maximizes the use of available data.

#### Additional comments

- The RCT was stopped due to practice changes, which can introduce bias. Early-stopped trials may overestimate the treatment effect or otherwise affect the interpretability of results.
- With a relatively small sample size and potential imbalance in covariates, randomization alone might not ensure balance (even if p-values are > 0.05). Hence, adjusting for known confounders is critical.
- Be wary of exaggerated findings, as smaller studies are more prone to exaggeration.
  - Known as a Type M (magnitude) error. In other words, a finding must be large enough to exceed the statistical significance threshold despite wide confidence intervals, which systematically inflates the estimated effect size. Consequently, although we observed a strong effect, its true magnitude may be substantially lower than our point estimate suggests.[1]

#### References

Gelman, A., & Carlin, J. (2014). Beyond Power Calculations: Assessing Type S (Sign) and Type M (Magnitude) Errors. Perspectives on Psychological Science, 9(6), 641-651. https://doi.org/10.1177/1745691614551642

René-Sosata Bun, Jordan Scheer, Sylvie Guillo, Florence Tubach, Agnès Dechartres, Meta-analyses frequently pooled different study types together: a meta-epidemiological study, Journal of Clinical Epidemiology, Volume 118, 2020, Pages 18-28, ISSN 0895-4356, https://doi.org/10.1016/j.jclinepi.2019.10.013.

Sarri G, Patorno E, Yuan H, et alFramework for the synthesis of non-randomised studies and randomised controlled trials: a guidance on conducting a systematic review and meta-analysis for healthcare decision makingBMJ Evidence-Based Medicine 2022;27:109-119.

Shrier I, Boivin JF, Steele RJ, Platt RW, Furlan A, Kakuma R, Brophy J, Rossignol M. Should meta-analyses of interventions include observational studies in addition to randomized controlled trials? A critical examination of underlying principles. Am J Epidemiol. 2007 Nov 15;166(10):1203-9. doi: 10.1093/aje/kwm189. Epub 2007 Aug 21. PMID: 17712019.

# Additional Exclusion Criteria



# Tables

# **Baseline Characteristics**

Table 1a: Baseline demographics, randomized patients

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| | | (N=16) | (N=30) | |
| Gender: Male Days from surgery to last follow-up | 46<br>46 | 6/16 (37.50) | 16/30 (53.33) | X <sup>2</sup> <sub>1</sub> =1.05, P=0.31 <sup>2</sup><br>F <sub>1,44</sub> =5.51, P=0.02 <sup>3</sup> |
| N | 40 | 16 | 30 | F1,44=3.31, F=0.02 |
| Median (interquartile range) | | 1157.50 (727.67 – 1672.42) | 544.00 (140.92-1226.92) | |
| Range | | 76.00-3100.00 | 0.00-2157.00 | |
| Mean±SD | | 1191.38±774.56 | 710.13±632.56 | |
| Age | 46 | | | F <sub>1.44</sub> =2.51. P=0.12 <sup>3</sup> |
| N<br>Madian (interpretal property) | | 16 | 30 | |
| Median (interquartile range) | | 60.00 (55.83 – 68.58) | 57.00 (43.00 – 62.08) | |
| Range | | 27.00 — 75.00 | 20.00-73.00 | |
| Mean±SD<br>Body mass index | 46 | 59.25±13.79 | 53.57±13.50 | F <sub>1,44</sub> =1.23, P=0.27 <sup>3</sup> |
| N | 40 | 16 | 30 | 11,44-1.25, 1-0.27 |
| Median (interquartile range) | | 29.61 (26.79 – 33.45) | 33.10 (26.46-37.38) | |
| Range | | 21.22-40.21 | 20.91-42.16 | |
| Mean±SD | | 30.14±5.03 | 32.21±6.21 | |
| BMI >30kg/m2 : Yes | 46 | 8/16 (50.00) | 18/30 (60.00) | $X_{21}^{2}=0.42$ . P=0.51 <sup>2</sup> |
| Diabetes: Yes | 46 | 7/16 (43.75) | 7/30 (23.33) | $X^2_{1}=2.05$ , $P=0.15^2$ |
| Hypertension: Yes | 46 | 7/16 (43.75) | 14/30 (46.67) | $X^2_1=0.04$ , P=0.85 <sup>2</sup> |
| COPD: Yes | 46 | 5/16 (31.25) | 5/30 (16.67) | $X^{2}_{1}=1.30$ , $P=0.25^{2}$ |
| Immunosuppression : Yes Primary hernia diagnosis : Yes | 46<br>46 | 2/16 (12.50)<br>14/16 (87.50) | 10/30 (33.33)<br>28/30 (93.33) | X <sup>2</sup> <sub>1</sub> =2.35, P=0.13 <sup>2</sup><br>X <sup>2</sup> <sub>1</sub> =0.45, P=0.50 <sup>2</sup> |
| Previous repair : Yes | 46 | 11/16 (68.75) | 20/30 (93.33) | $X^{1}=0.45, P=0.50$<br>$X^{2}_{1}=0.02, P=0.89^{2}$ |
| Number of prior hernia repairs | 46 | | | F <sub>1,44</sub> =1.93, P=0.17 <sup>3</sup> |
| N | | 16 | 30 | |
| Median (interquartile range) | | 2.50 (0.00-4.58) | 1.00 (0.00-2.00) | |
| Range | | 0.00-9.00 | 0.00-6.00 | |
| Mean±SD<br>History of mesh repair : Yes | 46 | 2.69±2.73<br>12/16 (75.00) | 1.43±1.61<br>17/30 (56.67) | X <sup>2</sup> <sub>1</sub> =1.51, P=0.22 <sup>2</sup> |
| , I | | 12/10 (73.00) | 17/30 (30.07) | |
| Hernia width | 41 | 17 | 0.5 | F <sub>1,39</sub> =2.14, P=0.15 <sup>3</sup> |
| N<br>Median (interquartile range) | | 16<br>15.80 (9.95—18.71) | 25<br>12.60 (9.20—14.80) | |
| Range | | 2.10—30.30 | 2.20—22.20 | |
| Mean±SD | | 14.91±7.41 | 11.67±5.48 | |
| Hernia width (imputed) | 46 | | | F <sub>1,44</sub> =0.68, P=0.41 <sup>3</sup> |
| N | | 16 | 30 | |
| Median (interquartile range) | | 15.80 (9.95—18.71) | 12.90 (9.48—18.65) | |
| Range<br>Mean±SD | | 2.10-30.30<br>14.91±7.41 | 2.20-30.00<br>13.06±6.46 | |
| | | 14.7127.41 | 15.0020.40 | - 0.10 P.0==2 |
| Hernia length | 41 | 16 | 25 | F <sub>1,39</sub> =0.10, P=0.75 <sup>3</sup> |
| N<br>Median (interquartile range) | | 16<br>16.60 (9.84—20.00) | 25<br>11.80 (8.20—21.60) | |
| Range | | 2.30—28.00 | 3.50-27.70 | |
| Mean±SD | | 15.30±6.90 | 14.20±7.89 | |
| Hernia length (imputed) | 46 | | | F <sub>1,44</sub> =0.01, P=0.93 <sup>3</sup> |
| N | | 16 | 30 | |
| Median (interquartile range) | | 16.60 (9.84—20.00) | 16.25 (9.00—21.41) | |
| Range<br>Mean±SD | | 2.30-28.00<br>15.30±6.90 | 3.50-27.70<br>15.05±7.49 | |
| | 4.4 | 10.0010.70 | 10.0027.17 | E 100 D002 |
| Hernia area | 41 | 16 | 25 | F <sub>1,39</sub> =1.33, P=0.26 <sup>3</sup> |
| N<br>Median (interquartile range) | | 16<br>275.97 (96.08—354.27) | 25<br>153.40 (45.61—301.15) | |
| Range | | 8.61—700.00 | 7.70 — 545.69 | |
| Mean±SD | | 265.97±200.88 | 195.61±157.45 | |
| Total OR time (min) | 43 | | | F <sub>1,41</sub> =0.29, P=0.59 <sup>3</sup> |
| N | | 14 | 29 | |
| Median (interquartile range) | | 471.50 (443.50—483.58) | 417.00 (336.33 – 547.67) | |
| Range<br>Mean±SD | | 292.00 — 560.00<br>462.57±58.22 | 212.00 — 838.00<br>451.17±142.81 | |
| | | 102.07 ±00.22 | 101,17 ±174,01 | |
| ASA class | 46 | 2/17 (10 55) | 2/20 /10 00) | $X^2_2=2.21$ , P=0.33 <sup>2</sup> |
| 2 | | 3/16 (18.75) | 3/30 (10.00) | |
| J | | 13/16 (81.25) | 24/30 (80.00) | |

Table 1a: Baseline demographics, randomized patients (continued)

| Variables | N | Strattice | XenMatrix | Test Statistic |
|-----------|---|-------------|--------------|----------------|
| 4 | | 0/16 (0.00) | 3/30 (10.00) | |

#### Note.

N is the number of non-missing value. 1 Kruskal-Wallis. 2 Pearson. 3 Wilcoxon. Stat, P is the test statistic and p-value. cata = check all that apply

Table 1b: Baseline demographics, observational patients

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| Gender: Male | 20<br>20 | (N=12)<br>6/12 (50.00) | (N=8)<br>3/8 (37.50) | X <sup>2</sup> <sub>1</sub> =0.30, P=0.58 <sup>2</sup><br>F <sub>1,18</sub> =1.18, P=0.29 <sup>3</sup> |
| Days from surgery to last follow-up N | 20 | 12 | 8 | F1,18=1.16, F=0.29 |
| Median (interquartile range) | | 311.50 (93.67—469.17) | 570.50 (156.75—1293.50) | |
| Range<br>Mean±SD | | 54.00 — 855.00<br>327.08±266.89 | 64.00 — 1751.00<br>715.38±669.49 | |
| Age<br>N | 20 | 12 | 8 | F <sub>1,18</sub> =0.01, P=0.94 <sup>3</sup> |
| Median (interquartile range) | | 55.00 (49.42 – 60.58) | 57.50 (35.33 – 67.58) | |
| Range | | 32.00-70.00 | 30.00-73.00 | |
| Mean±SD<br>Body mass index | 20 | 54.75±10.16 | 53.12±17.01 | F <sub>1,18</sub> =2.30, P=0.15 <sup>3</sup> |
| N<br>Median (interquartile range) | | 12<br>36.48 (32.12—38.26) | 8<br>32.97 (25.34—35.71) | |
| Range<br>Mean±SD | | 24.17—47.60<br>35.59±6.02 | 21.49 – 39.67<br>31.23±6.49 | |
| BMI >30kg/m2 : Yes<br>Diabetes : Yes | 20<br>20 | 10/12 (83.33)<br>2/12 (16.67) | 5/8 (62.50)<br>0/8 (0.00) | X <sup>2</sup> <sub>1</sub> =1.11. P=0.29 <sup>2</sup><br>X <sup>2</sup> <sub>1</sub> =1.48, P=0.22 <sup>2</sup> |
| Hypertension: Yes | 20 | 7/12 (58.33) | 2/8 (25.00) | $X^2_1=2.15$ , $P=0.14^2$ |
| COPD : Yes<br>Immunosuppression : Yes | 20<br>20 | 1/12 (8.33)<br>4/12 (33.33) | 1/8 (12.50)<br>0/8 (0.00) | X <sup>2</sup> <sub>1</sub> =0.09, P=0.76 <sup>2</sup><br>X <sup>2</sup> <sub>1</sub> =3.33, P=0.07 <sup>2</sup> |
| Primary hernia diagnosis : Yes<br>Previous repair : Yes | 20<br>20 | 4/12 (33.33)<br>7/12 (58.33) | 7/8 (87.50)<br>3/8 (37.50) | X <sup>2</sup> <sub>1</sub> =5.69, P=0.02 <sup>2</sup><br>X <sup>2</sup> <sub>1</sub> =0.83, P=0.36 <sup>2</sup> |
| Number of prior hernia repairs | 20 | | | F <sub>1,18</sub> =0.33, P=0.57 <sup>3</sup> |
| N | | 12 | 8 | |
| Median (interquartile range)<br>Range | | 1.00 (0.00—1.58)<br>0.00—9.00 | 0.00 (0.00—2.17)<br>0.00—6.00 | |
| Mean±SD | 20 | 1.50±2.54 | 1.25±2.19 | V <sup>2</sup> 0.20 D.050 <sup>2</sup> |
| History of mesh repair : Yes | 20 | 6/12 (50.00) | 3/8 (37.50) | $X^{2}_{1}=0.30$ , $P=0.58^{2}$ |
| Hernia width<br>N | 19 | 11 | 8 | $F_{1,17}=5.27$ , $P=0.03^3$ |
| Median (interquartile range)<br>Range | | 11.70 (9.75—16.47)<br>2.80—30.00 | 16.50 (15.27—19.93)<br>15.00—22.50 | |
| Mean±SD | | 13.23±7.78 | 17.54±2.94 | _ |
| Hernia width (imputed) | 20 | 10 | 0 | F <sub>1,18</sub> =2.89, P=0.11 <sup>3</sup> |
| N<br>Median (interquartile range) | | 12<br>12.45 (9.82—20.15) | 8<br>16.50 (15.27—19.93) | |
| Range | | 2.80 – 30.00 | 15.00 — 22.50 | |
| Mean±SD | 40 | 14.62±8.86 | 17.54±2.94 | E 0.04 D.0013 |
| Hernia length<br>N | 19 | 11 | 8 | F <sub>1,17</sub> =0.01, P=0.91 <sup>3</sup> |
| Median (interquartile range)<br>Range | | 22.50 (20.10—25.08)<br>2.40—32.70 | 22.35 (19.17—27.41)<br>13.50—30.00 | |
| Mean±SD | | 20.27±9.01 | 22.61±5.47 | - |
| Hernia length (imputed) N | 20 | 12 | 8 | F <sub>1,18</sub> =0.07, P=0.80 <sup>3</sup> |
| Median (interquartile range) | | 22.05 (20.00—24.91) | 22.35 (19.17—27.41) | |
| Range<br>Mean±SD | | 2.40 — 32.70<br>20.25±8.59 | 13.50 — 30.00<br>22.61±5.47 | |
| Hernia area | 19 | 11 | 0 | F <sub>1,17</sub> =2.69, P=0.12 <sup>3</sup> |
| N<br>Median (interquartile range) | | 11<br>284.28 (231.27—422.23) | 8<br>362.85 (322.09—467.22) | |
| Range Mean±SD | | 6.72 — 600.00<br>298.77±188.98 | 230.90 – 657.00<br>398.54±130.54 | |

Table 1b: Baseline demographics, observational patients (continued)

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| Total OR time (min) | 19 | | | F <sub>1,17</sub> =0.34, P=0.57 <sup>3</sup> |
| N | | 12 | 7 | |
| Median (interquartile range) | | 431.00 (383.17 - 540.58) | 551.00 (345.17-575.83) | |
| Range | | 310.00-696.00 | 289.00-1018.00 | |
| Mean±SD | | 465.08±117.42 | 538.86±240.86 | |
| ASA class | 20 | | | $X^2_2=3.59$ , P=0.17 <sup>2</sup> |
| 2 | | 1/12 (8.33) | 1/8 (12.50) | |
| 3 | | 11/12 (91.67) | 5/8 (62.50) | |
| 4 | | 0/12 (0.00) | 2/8 (25.00) | |

Note:

N is the number of non-missing value. 1 Kruskal-Wallis. 2 Pearson. 3 Wilcoxon.

Stat, P is the test statistic and p-value.

cata = check all that apply

# **Surgical Characteristics**

Table 2a: Surgical demographics, randomized patients

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| | | (N=16) | (N=30) | |
| Types of hernia diagnosis <sup>cata</sup> | | | | |
| Ventral hernia : Yes | 46 | 15/16 (93.75) | 28/30 (93.33) | $X^2_1=0.00$ , $P=0.96^2$ |
| Flank hernia : Yes | 46 | 0/16 (0.00) | 2/30 (6.67) | X <sup>2</sup> <sub>1</sub> =1.12, P=0.29 <sup>2</sup> |
| Parastomal hernia : Yes | 46 | 3/16 (18.75) | 3/30 (10.00) | $X^2_1=0.70$ , $P=0.40^2$ |
| Umbilical hernia : Yes | 46 | 0/16 (0.00) | 0/30 (0.00) | NA |
| Parastomal hernia : Yes | 46 | 3/16 (18.75) | 3/30 (10.00) | $X^2_1=0.70$ , P=0.40 <sup>2</sup> |
| CDC wound class | 46 | | | $X^2_3=3.08$ , P=0.38 <sup>2</sup> |
| 1 | | 7/16 (43.75) | 17/30 (56.67) | |
| 2 | | 5/16 (31.25) | 4/30 (13.33) | |
| 3 | | 2/16 (12.50) | 2/30 (6.67) | |
| 4 | | 2/16 (12.50) | 7/30 (23.33) | |
| VHWG grade | 46 | | | $X^2_3=3.46$ , P=0.33 <sup>2</sup> |
| 1 | | 1/16 (6.25) | 1/30 (3.33) | |
| 2 | | 2/16 (12.50) | 9/30 (30.00) | |
| 3 | | 11/16 (68.75) | 13/30 (43.33) | |
| 4 | | 2/16 (12.50) | 7/30 (23.33) | |
| Kanters grade | 46 | | | $X^2 = 1.12$ . $P = 0.57^2$ |
| 1 | | 1/16 (6.25) | 1/30 (3.33) | |
| 2 | | 6/16 (37.50) | 16/30 (53.33) | |
| 3 | | 9/16 (56.25) | 13/30 (43.33) | |
| Primary fascial repair: Yes | 46 | 14/16 (87.50) | 22/30 (73.33) | $X^2_1=1.23$ . P=0.27 <sup>2</sup> |
| Unilateral component separation : Yes | 46 | 2/16 (12.50) | 2/30 (6.67) | $X^2_1=0.45$ , $P=0.50^2$ |
| Bilateral component separation : Yes | 46 | 8/16 (50.00) | 17/30 (56.67) | $X^2_{1}=0.19$ . P=0.67 <sup>2</sup> |
| Bridged repair : Yes | 46 | 2/16 (12.50) | 6/30 (20.00) | $X^2_1=0.41$ , $P=0.52^2$ |
| Mesh position <sup>cata</sup> | | | | 2 |
| Onlay mesh placement : Yes | 46 | 0/16 (0.00) | 3/30 (10.00) | $X^2_1=1.71$ , $P=0.19^2$ |
| Underlay mesh placement : Yes | 46 | 12/16 (75.00) | 24/30 (80.00) | $X^{2}_{1}=0.15$ , P=0.70 <sup>2</sup> |
| Inlay mesh placement : Yes<br>Sublay mesh placement : Yes | 46<br>46 | 0/16 (0.00)<br>4/16 (25.00) | 2/30 (6.67)<br>8/30 (26.67) | $X^{2}_{1}=1.12$ , $P=0.29^{2}$<br>$X^{2}_{1}=0.02$ , $P=0.90^{2}$ |
| Subiay mesh piacement: Tes | 40 | 4/10 (23.00) | 0/30 (20.07) | ∧ 1-0.02, F=0.90 |

Note:

N is the number of non-missing value. 1 Kruskal-Wallis. 2 Pearson. 3 Wilcoxon.

Stat, P is the test statistic and p-value.

cata = check all that apply

Table 2b: Surgical demographics, observational patients

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| | | (N=12) | (N=8) | |
| Types of hernia diagnosis <sup>cata</sup> | | | | |
| Ventral hernia : Yes | 20 | 11/12 (91.67) | 7/8 (87.50) | $X^2_1=0.09$ , P=0.76 <sup>2</sup> |
| Flank hernia: Yes | 20 | 2/12 (16.67) | 1/8 (12.50) | $X^2_1=0.07$ , P=0.80 <sup>2</sup> |
| Parastomal hernia : Yes | 20 | 4/12 (33.33) | 0/8 (0.00) | $X^2_1=3.33$ , $P=0.07^2$ |

Table 2b: Surgical demographics, observational patients (continued)

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| Umbilical hernia : Yes | 20 | 0/12 (0.00) | 0/8 (0.00) | NA |
| Parastomal hernia: Yes | 20 | 4/12 (33.33) | 0/8 (0.00) | $X^2_1=3.33$ , $P=0.07^2$ |
| CDC wound class | 20 | | ` , | $X^2_3=3.64$ . P=0.30 <sup>2</sup> |
| 1 | | 6/12 (50.00) | 5/8 (62.50) | |
| 2 | | 3/12 (25.00) | 2/8 (25.00) | |
| 3 | | 0/12 (0.00) | 1/8 (12.50) | |
| 4 | | 3/12 (25.00) | 0/8 (0.00) | |
| VHWG grade | 20 | | | $X^2_3=4.49$ , $P=0.21^2$ |
| 1 | | 0/12 (0.00) | 1/8 (12.50) | |
| 2 | | 6/12 (50.00) | 2/8 (25.00) | |
| 3 | | 4/12 (33.33) | 5/8 (62.50) | |
| 4 | | 2/12 (16.67) | 0/8 (0.00) | |
| Kanters grade | 20 | | | $X^2_{1}=0.83$ . P=0.36 <sup>2</sup> |
| 1 | | 0/12 (0.00) | 0/8 (0.00) | |
| 2 | | 5/12 (41.67) | 5/8 (62.50) | |
| 3 | | 7/12 (58.33) | 3/8 (37.50) | |
| Primary fascial repair : Yes | 19 | 9/12 (75.00) | 6/7 (85.71) | $X^2_1=0.31$ , $P=0.58^2$ |
| Unilateral component separation: Yes | 20 | 1/12 (8.33) | 0/8 (0.00) | $X^2_1=0.70$ , $P=0.40^2$ |
| Bilateral component separation: Yes | 20 | 4/12 (33.33) | 7/8 (87.50) | $X_{1}^{2}=5.69$ . P=0.02 <sup>2</sup> |
| Bridged repair : Yes | 19 | 4/12 (33.33) | 1/7 (14.29) | $X^2_1=0.83$ , $P=0.36^2$ |
| Mesh position <sup>cata</sup> | | | | |
| Onlay mesh placement : Yes | 20 | 0/12 (0.00) | 0/8 (0.00) | NA |
| Underlay mesh placement: Yes | 20 | 12/12 (100.00) | 6/8 (75.00) | $X^2_1=3.33$ , $P=0.07^2$ |
| Inlay mesh placement : Yes | 20 | 1/12 (8.33) | 1/8 (12.50) | $X^2_1=0.09$ , $P=0.76^2$ |
| Sublay mesh placement: Yes | 20 | 0/12 (0.00) | 2/8 (25.00) | $X^2_{1}=3.33$ , P=0.07 <sup>2</sup> |

N is the number of non-missing value. 1 Kruskal-Wallis. 2 Pearson. 3 Wilcoxon.

Stat, P is the test statistic and p-value.

cata = check all that apply

## 6-week Outcomes

Table 3a: 6-week outcomes, randomized patients

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| | | (N=16) | (N=30) | |
| Bulge · Yes | 46 | 0/16 (0.00) | 0/30 (0.00) | NA |
| Bulge : Yes<br>Recurrence : Yes | 46 | 0/16 (0.00) | 0/30 (0.00)<br>0/30 (0.00) | ŇÄ |
| SSO within 6 weeks: Yes | 46 | 1/16 (6.25) | 11/30 (36.67) | $X^2_1=5.01$ , P=0.03 <sup>2</sup> |
| SSO Type (cata) | | | | |
| | 4.0 | 0.44.6.40.000 | 1 (00 (0.00) | 3/2 0 == D 0 4/2 |
| Skin necrosis: Yes | 46 | 0/16 (0.00) | 1/30 (3.33) | $X^2_1=0.55$ , $P=0.46^2$ |
| Enterocutaneous fistula : Yes | 46 | 0/16 (0.00) | 2/30 (6.67) | $X^{2}_{1}=1.12$ , P=0.29 <sup>2</sup> |
| Dehiscence: Yes | 46 | 0/16 (0.00) | 1/30 (3.33) | $X^{2}_{1}=0.55$ , P=0.46 <sup>2</sup> |
| Seroma: Yes | 46 | 0/16 (0.00) | 2/30 (6.67) | $X^2_1=1.12$ , $P=0.29^2$ |
| Hematoma : Yes | 46 | 0/16 (0.00) | 0/30 (0.00) | NA |
| | | , | , , , | |
| Infection: Yes | 46 | 1/16 (6.25) | 10/30 (33.33) | $X^2_1=4.21$ , $P=0.04^2$ |
| Mesh infection: Yes | 46 | 0/16 (0.00) | 3/30 (10.00) | X <sup>2</sup> <sub>1</sub> =1.71, P=0.19 <sup>2</sup> |

N is the number of non-missing value. 1 Kruskal-Wallis. 2 Pearson. 3 Wilcoxon.

Stat, P is the test statistic and p-value.

cata = check all that apply

Table 3b: 6-week outcomes, observational patients

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| | | (N=12) | (N=8) | |
| Bulge · Yes<br>Recurrence : Yes<br>SSO within 6 weeks : Yes<br>SSO Type (cata) | 20<br>20<br>20 | 0/12 (0.00)<br>1/12 (8.33)<br>4/12 (33.33) | 0/8 (0.00)<br>0/8 (0.00)<br>4/8 (50.00) | NA<br>X <sup>2</sup> <sub>1</sub> =0.70, P=0.40 <sup>2</sup><br>X <sup>2</sup> <sub>1</sub> =0.56, P=0.46 <sup>2</sup> |
| Skin necrosis : Yes<br>Enterocutaneous fistula : Yes | 20<br>20 | 0/12 (0.00)<br>2/12 (16.67) | 1/8 (12.50)<br>0/8 (0.00) | X <sup>2</sup> <sub>1</sub> =1.58, P=0.21 <sup>2</sup><br>X <sup>2</sup> <sub>1</sub> =1.48, P=0.22 <sup>2</sup> |

Table 3b: 6-week outcomes, observational patients (continued)

| Variables | N | Strattice | XenMatrix | Test Statistic |
|---|---|---|---|---|
| Dehiscence: Yes | 20 | 2/12 (16.67) | 0/8 (0.00) | X <sup>2</sup> <sub>1</sub> =1.48, P=0.22 <sup>2</sup> |
| Seroma: Yes | 20 | 1/12 (8.33) | 0/8 (0.00) | $X^2_1=0.70$ , $P=0.40^2$ |
| Hematoma : Yes | 20 | 0/12 (0.00) | 0/8 (0.00) | NA |
| Infection: Yes | 20 | 1/12 (8.33) | 3/8 (37.50) | $X^2_1=2.55$ , P=0.11 <sup>2</sup> |
| Mesh infection: Yes | 19 | 0/11 (0.00) | 0/8 (0.00) | NA |

#### Note:

N is the number of non-missing value. 1 Kruskal-Wallis. 2 Pearson. 3 Wilcoxon. Stat, P is the test statistic and p-value.

cata = check all that apply

## **Results**

## **Executive Summary**

#### Unadjusted Random Effects Meta-Analysis (Simple Logistic Regression):

Effect Estimate (Odds Ratio): 3.718 (0.897, 15.404)

Significance: The pooled estimate was not statistically significant.

Heterogeneity:

 $I^2$  (total heterogeneity / total variability): 3.29%  $H^2$  (total variability / sampling variability): 1.03

Test for Heterogeneity:

Q(df = 1) = 1.0340, p-val = 0.3092

There appears to be minimal variability between the two studies. The  $I^2$  value of 3.29% indicates that nearly all of the total variation can be explained by chance rather than true heterogeneity, and an  $H^2$  of 1.03 reflects low excess variability. The Q test (Q = 1.034, p = 0.3092) is nonsignificant, confirming that there is no strong evidence of meaningful heterogeneity.

#### Adjusted Random Effects Meta-Analysis (Multivariable Logistic Regression):

Effect Estimate (Odds Ratio): 12.476 (1.745, 89.199)

Significance: The pooled estimate was statistically significant.

Heterogeneity:

 $I^2$  (total heterogeneity / total variability): 0.00%  $H^2$  (total variability / sampling variability): 1.00

Test for Heterogeneity: Q(df = 1) = 0.2830, p-val = 0.5947

There is effectively no evidence of meaningful heterogeneity between the RCT and the observational study, provided by  $0.00\% I^2$  value. Similarly,  $H^2 = 1.00$  supports the absence of excess variability beyond what would be expected by sampling error alone. Finally, the Q test (Q = 0.2830, p = 0.5947) is non-significant, confirming that the studies are consistent and do not exhibit statistically detectable heterogeneity.

When covariates were included in the model, a previously non-significant association between the exposure and outcome became statistically significant. This shift suggests that the unadjusted analysis may have been confounded—i.e., certain variables were masking or biasing the relationship.

#### Note

Be wary of exaggerated findings, as smaller studies are more prone to exaggeration. This is known as a Type M (magnitude) error. In other words, a finding must be large enough to exceed the statistical significance threshold despite wide confidence intervals, which systematically inflates the estimated effect size. Consequently, although we observed a strong effect, its true magnitude may be substantially lower than our point estimate suggests.

Gelman, A., & Carlin, J. (2014). Beyond Power Calculations: Assessing Type S (Sign) and Type M (Magnitude) Errors. Perspectives on Psychological Science, 9(6), 641-651.

# Random Effects Meta-Analysis: Simple Logistic Regression

Simple logistic regression = logistic regression with no adjustment for confounders

Random Effects Meta-Analysis: Simple Logistic Regression

| Study | Estimate (log OR) | 95% CI (log OR) | Estimate (OR) | 95% CI (OR) | P-value |
|---|---|---|---|---|---|
| Randomized | 2.162 | (0.365, 5.123) | 8.684 | (1.441, 167.853) | 0.049 |
| Observational | 0.693 | (-1.143, 2.597) | 2.000 | (0.319, 13.423) | 0.459 |
| RE Meta-Analysis | 1.313 | (-0.108, 2.735) | 3.718 | (0.897, 15.404) | 0.070 |

Forest Plot: Log Odds Scale





# Random Effects Meta-Analysis: Multivariable logistic regression

Random Effects Meta-Analysis: Multivariable Logistic Regression

| Study | Estimate (log OR) | 95% CI (log OR) | Estimate (OR) | 95% CI (OR) | P-value |
|---|---|---|---|---|---|
| Randomized | 2.968 | (0.815, 6.261) | 19.458 | (2.258, 523.717) | 0.023 |
| Observational | 1.882 | (-0.898, 5.783) | 6.569 | (0.407, 324.629) | 0.230 |
| RE Meta-Analysis | 2.524 | (0.557, 4.491) | 12.476 | (1.745, 89.199) | 0.012 |

# Log Odds Scale





# **FAO**

#### Q: What is overfitting?

A: Overfitting in regression happens when a model is too complex, often due to too many parameters relative to a small sample size, causing it to capture noise rather than the true data pattern. With limited data, the model lacks sufficient information to generalize well, leading to poor performance on new data because it is overly tailored to the specific quirks of the training set.

#### Q: What is a chunk (or composite) test?

A: A chunk or composite hypothesis test is often used for categorical variables to assess whether the entire variable contributes significantly to the model, rather than just specific categories. By testing all categories together, this approach helps determine if the variable as a whole has an effect, rather than focusing on individual category differences alone.

#### Q: What can I say when I have a large p-value?

A. This is a friendly reminder that absence of evidence does not mean evidence of absence. A large p-value doesn't prove there is no effect; it simply indicates that we don't have strong evidence to detect a difference. Instead of incorrectly concluding "there were no differences," it's more accurate to say, "there was no evidence of a difference." Additionally, you can use the confidence interval to provide more context. For example, if comparing complication rates, and the confidence interval suggests the difference could be as much as ±5 percentage points, you might say: "If there is a difference between procedure A and procedure B, it is likely no larger than 5 percentage points." Similarly, for odds ratios, if the confidence interval includes a range up to 2, you could say, "There may be at most a 100% increase in odds or up to a 50% decrease in odds." This acknowledges uncertainty without overinterpreting the results.

Answer generously borrowed and adapted from this blog post(link) by Thomas Stewart, PhD.

Also see this article for explanation of interpretation of evidence and suggestions about communicating levels of evidence.

#### Q. What is validation and optimism-corrected statistics?

A. When a model is fit to a dataset, it tends to perform better on that dataset than it would on new, unseen data, leading to overly optimistic predictions and performance statistics. To adjust for this, techniques like cross-validation or bootstrapping are used to correct for this optimism, producing "optimism-corrected" statistics, which provide a more realistic estimate of the model's performance on future data. These corrections help ensure that the model's results are not overly tailored to the training data and are more generalizable.

#### Q. What are Brier scores (B)?

A. The Brier score measures how well a model predicts binary or categorical outcomes by calculating the mean squared difference between the predicted probabilities and the actual outcomes. It ranges from 0 to 1, with lower scores indicating better predictive accuracy and calibration. A Brier score closer to 0 suggests that the model's predicted probabilities align well with the observed outcomes, making it a useful metric for evaluating the accuracy of probabilistic predictions.

#### Q. What is the g-index (g)?

A. The g-index measures the ability of a model to discriminate between outcomes based on the Gini mean difference, reflecting the typical difference between predictions for any two randomly selected individuals. In essence, a higher g-index indicates better discrimination, meaning the model provides a wider range of predictions that can distinguish between individuals more effectively. For example, in a time-to-event analysis, a larger g-index suggests that the model can predict meaningful differences in survival times or hazard rates between patients.

For time-to-event outcomes: A higher g-index indicates larger differences in predicted log relative hazards between patients, which implies better discrimination. For binary/ordinal outcomes: The g-index reflects the typical log odds ratio between predictions for any two patients, meaning how much their odds of an outcome differ. For continuous outcomes: The g-index represents the typical difference in predicted values, showing how far apart predictions are for different patients. Overall, a higher g-index means the model is better at distinguishing between individuals based on their predicted outcomes.

Here are improved explanations for each of your questions:

#### Q. What is validation and optimism-corrected statistics?

A. When a model is fit to a dataset, it tends to perform better on that dataset than it would on new, unseen data, leading to overly optimistic predictions and performance statistics. To adjust for this, techniques like cross-validation or bootstrapping are used to correct for this optimism, producing "optimism-corrected" statistics, which provide a more realistic estimate of the model's performance on future data. These corrections help ensure that the model's results are not overly tailored to the training data and are more generalizable.

#### Q. What are Brier scores (B)?

A. The Brier score measures how well a model predicts binary or categorical outcomes by calculating the mean squared difference between the predicted probabilities and the actual outcomes. It ranges from 0 to 1, with lower scores indicating better predictive accuracy and calibration. A Brier score closer to 0 suggests that the model's predicted probabilities align well with the observed outcomes, making it a useful metric for evaluating the accuracy of probabilistic predictions.

#### Q. What is the g-index (g)?

A. The g-index measures the ability of a model to discriminate between outcomes based on the Gini mean difference, reflecting the typical difference between predictions for any two randomly selected individuals. In essence, a higher g-index indicates better discrimination, meaning the model provides a wider range of predictions that can distinguish between individuals more effectively. For example, in a time-to-event analysis, a larger g-index suggests that the model can predict meaningful differences in survival times or hazard rates between patients.

For time-to-event outcomes: A higher g-index indicates larger differences in predicted log relative hazards between patients, which implies better discrimination. For binary/ordinal outcomes: The g-index reflects the typical log odds ratio between predictions for any two patients, meaning how much their odds of an outcome differ. For continuous outcomes: The g-index represents the typical difference in predicted values, showing how far apart predictions are for different patients. Overall, a higher g-index means the model is better at distinguishing between individuals based on their predicted outcomes.

g is on the original scale gr is on the ratio scale (e.g. odds/hazard) gp is on the probability or risk scale

#### Q. What is DXY?

A. Dxy, or Somers' Dxy, is a statistic used to measure a model's discrimination ability, which refers to how well the model can distinguish between different outcomes. Dxy ranges from -1 to 1, with 1 indicating perfect discrimination and 0 indicating no better than random guessing. For binary outcomes, Dxy is related to the concordance index (c-index) and can be expressed as Dxy = 2 \* (c-index - 0.5). In time-to-event models, Dxy represents the rank correlation between the predicted log relative hazard and observed survival times, similar to a rank-based R2. Higher Dxy values indicate that the model does a better job at ranking individuals according to their predicted outcomes.

#### For example:

Dxy = 0.5 means 75% of pairs are concordant (the predictions are in the correct order), and 25% are discordant. Dxy = 0.2 means 60% of pairs are concordant, and 40% are discordant. According to Dr. Frank Harrell, there are no universally "acceptable" values for Dxy, as the significance depends on the difficulty of predicting the specific outcome (e.g., lower values may still be informative for difficult-to-predict outcomes like mortality).

#### Q. What is a restricted cubic spline? What are knots?

A. Restricted cubic splines are a flexible tool used in statistical models to better capture non-linear relationships between a continuous variable and an outcome. Instead of assuming a straight-line relationship, restricted cubic splines break the data into sections at specific points, called "knots," and fit smooth curves between them. The "restricted" part means the curves become straight lines at the ends, ensuring the model doesn't overreact to extreme values. This method helps create a smoother, more realistic fit to the data without making the model too complicated or unstable, making it useful when simple linear relationships aren't sufficient.

#### Q. What is a tipping point analysis?

A. A tipping point analysis is a type of sensitivity analysis used to assess how robust the results of a study are to potential changes or assumptions, especially in the presence of missing data or uncertain parameters. It identifies the point at which the study's conclusions would change if certain assumptions or values were adjusted. In the context of missing data, for example, tipping point analysis can determine how much the imputed or missing data would need to shift in order to alter the outcome of the analysis. This helps evaluate the stability of the results and the impact of potential biases on the conclusions.

# Q. What are the benefits of adding the propensity score as a covariate when there aren't enough events to include multiple covariates directly?

A. When you don't have enough events to directly include multiple covariates in a model, adding the propensity score as a covariate offers several benefits. It reduces dimensionality by summarizing multiple covariates into a single variable, improving model stability and avoiding overfitting. This approach efficiently adjusts for confounders without the need for a large number of parameters, maintaining statistical power and reducing bias in small sample settings. Additionally, it helps avoid multicollinearity and provides flexibility across different types of models, making it a valuable tool when dealing with sparse data.

Reference: Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID: 21818162; PMCID: PMC3144483.

## R Session info

```
## R version 4.4.1 (2024-06-14)
## Platform: x86_64-apple-darwin20
## Running under: macOS 15.3
##
## Matrix products: default
## BLAS: /Library/Frameworks/R.framework/Versions/4.4-x86_64/Resources/lib/libRblas.0.dylib
## LAPACK: /Library/Frameworks/R.framework/Versions/4.4-x86 64/Resources/lib/libRlapack.dylib;
                                                                                                     LAPACK version
##
## locale:
## [1] en_US.UTF-8/en_US.UTF-8/en_US.UTF-8/en_US.UTF-8
## time zone: America/New York
## tzcode source: internal
##
## attached base packages:
## [1] stats
                 graphics grDevices utils
                                                 datasets methods base
##
## other attached packages:
   [1] broom.helpers_1.17.0 broom_1.0.7
##
                                                    rms_7.0-0
##
   [4] Hmisc_5.2-2
                              tangram_0.8.2
                                                    magrittr_2.0.3
## [7] R6_2.5.1
                              ggplot2_3.5.1
                                                    janitor_2.2.1
## [10] dplyr_1.1.4
                              here_1.0.1
                                                    knitr_1.49
## [13] kableExtra_1.4.0
##
## loaded via a namespace (and not attached):
   [1] gtable_0.3.6
                            xfun 0.49
                                                htmlwidgets_1.6.4
                                                                    lattice 0.22-6
   [5] vctrs_0.6.5
                            tools_4.4.1
                                                                    sandwich_3.1-1
##
                                                generics_0.1.3
## [9] tibble_3.2.1
                            cluster_2.1.6
                                                pkgconfig_2.0.3
                                                                    Matrix_1.7-0
## [13] data.table_1.16.4
                            checkmate 2.3.2
                                                lifecycle_1.0.4
                                                                    compiler 4.4.1
## [17] stringr_1.5.1
                            MatrixModels 0.5-3
                                                munsell 0.5.1
                                                                    codetools_0.2-20
                                                                    htmltools\_0.5.8.1
## [21] snakecase_0.11.1
                            SparseM_1.84-2
                                                quantreg_6.00
## [25] yaml_2.3.10
                            htmlTable_2.4.3
                                                Formula_1.2-5
                                                                    tidyr_1.3.1
## [29] pillar_1.10.0
                            MASS_7.3-60.2
                                                rpart_4.1.23
                                                                    multcomp_1.4-28
                                                digest_0.6.37
## [33] nlme_3.1-164
                            tidyselect_1.2.1
                                                                    mvtnorm_1.3-3
## [37] polspline_1.1.25
                                                purrr_1.0.2
                                                                    splines 4.4.1
                            stringi_1.8.4
## [41] rprojroot_2.0.4
                            fastmap_1.2.0
                                                grid_4.4.1
                                                                    colorspace_2.1-1
## [45] cli_3.6.3
                            base64enc_0.1-3
                                                survival 3.6-4
                                                                    TH.data_1.1-3
## [49] foreign_0.8-86
                            withr_3.0.2
                                                scales_1.3.0
                                                                    backports_1.5.0
## [53] lubridate_1.9.4
                            timechange_0.3.0
                                                rmarkdown_2.29
                                                                    nnet_7.3-19
## [57] gridExtra_2.3
                            zoo_1.8-12
                                                evaluate_1.0.1
                                                                    viridisLite_0.4.2
## [61] rlang 1.1.4
                            glue 1.8.0
                                                xml2 1.3.6
                                                                    svglite_2.1.3
## [65] rstudioapi_0.17.1
                            systemfonts_1.1.0
## To cite R in publications use:
##
##
     R Core Team (2024). _R: A Language and Environment for Statistical
##
     Computing . R Foundation for Statistical Computing, Vienna, Austria.
##
     <a href="https://www.R-project.org/">https://www.R-project.org/>.</a>
##
## A BibTeX entry for LaTeX users is
##
##
     @Manual{,
##
       title = {R: A Language and Environment for Statistical Computing},
##
       author = {{R Core Team}},
##
       organization = {R Foundation for Statistical Computing},
##
       address = {Vienna, Austria},
##
       year = \{2024\},
##
       url = {https://www.R-project.org/},
##
##
```

## We have invested a lot of time and effort in creating R, please cite it ## when using it for data analysis. See also 'citation("pkgname")' for

## citing R packages.